CLINICAL TRIAL: NCT04431427
Title: Partially Covered Metal Stents Efficacy in the Biliary Drainage of Malignant Extra-hepatic Biliary Obstruction, a Multicentric Randomized Trial
Brief Title: Partially Covered Metal Stents Efficacy in Biliary Drainage of Malignant Extra-hepatic Biliary Obstruction
Acronym: METARSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Santi Mangiafico (Other)
Responsible Party: Sponsor-Investigator, Santi Mangiafico, Medical Doctor, Azienda Ospedaliero-Universitaria di Modena
Organization: Azienda Ospedaliero-Universitaria di Modena (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05.2020
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Biliary Obstruction
Keywords: Malignant biliary obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Partially Covered Metal Stent Arm (Active Comparator): The patients who had extra-hepatic malignant biliary obstruction will be enrolled in our study. Enrolled patient will be randomized to two group (uncovered metallic stent vs. partially covered metallic stent). After metallic biliary stent insertion, enrolled patients will be followed until bilirubin values will be under 2 mg/dl.
  Interventions: Device: Biliary drainage with PC-SEMS
- Uncovered Metal Stent Arm (Active Comparator): The patients who had extra-hepatic malignant biliary obstruction will be enrolled in our study. Enrolled patient will be randomized to two group (uncovered metallic stent vs. partially covered metallic stent). After metallic biliary stent insertion, enrolled patients will be followed until bilirubin values will be under 2 mg/dl.
  Interventions: Device: Biliary drainage with U-SEMS

INTERVENTIONS:
Device: Biliary drainage with PC-SEMS — partially covered metallic biliary stent insertion during ERCP
  Arms: Partially Covered Metal Stent Arm
Device: Biliary drainage with U-SEMS — Uncovered metallic biliary stent insertion during ERCP
  Arms: Uncovered Metal Stent Arm

SUMMARY:
Malignant obstructions of the bile duct are not rare. The most common and accepted method for biliary drainage is endoscopic stent placement. There are three types of metal stents: fully covered (FC), partially covered (PC) and uncovered (U). PC-SEMS have been recently introduced and compared to FC-SEMS they seem to have a lower risk of migration, although data in the literature are discordant. Therefore the investigators will randomize the participants with biliary obstruction in 2 groups according to the type of stent used: PC-SEMS or U-SEMS. After metallic biliary stent insertion, enrolled patients will be followed for 12 months.

DETAILED DESCRIPTION:
Malignant obstructions of the bile duct are generally caused by: adenocarcinoma of the Vater ampulla, pancreas head cancer, cholangiocarcinoma and external compression secondary to lymph node (LN) metastasis. The management of jaundice and cholangitis, as a result of bile stenosis, is crucial in this group of patients. The most common and accepted method for biliary drainage is endoscopic stent placement with plastic stents or self-expandable metal stents (SEMS). In recent times, the use of SEMS has become more common as it provides longer times of patency and a reduced risk of adverse events such as cholangitic episodes. There are three types of metal stents: fully covered (FC), partially covered (PC) and uncovered (U). PC-SEMS have been recently introduced and compared to FC-SEMS they seem to have a lower risk of migration, however different randomized and non-randomized studies have compared the outcome of U-SEMS vs FC-SEMS with between uncovered and covered stents have produced different results regarding the cumulative patency of stents and endoscopic re-intervention rates. To date, there are few and discordant prospective data on the outcomes of PC-SEMS use in malignant biliary obstructions.

Therefore, the investigators will randomize the participants with biliary obstruction in 2 groups according to the type of stent used: PC-SEMS or U-SEMS (T0 timing).

Then the participants will be followed for total period of 12 months. 2 different timings of follow-up will be considered:

- T1: it will start after stent insertion. The biliary drainage will be considered effective, according to the European guidelines, when the bilirubin values will be < or = 2 mg/dl for a period of at least 6 weeks if the initial bilirubin values were higher than 10 mg/dl or 3 weeks if at the beginning were lower than 10 mg/dl; After this first phase, all the enrolled patients will be divided in 2 groups according to their "fitness" for chemiotherapy: FIT and UNFIT Group.

FIT group: blood test (including total bilirubin, gamma-GT) will be done for follow-up study once every three months.

UNFIT Group: blood test (including total bilirubin, gamma-GT) will be done for follow-up study after 3, 9 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

•The patients who had malignant biliary obstruction with a estimated survival >4 months

Exclusion Criteria:

* The patients who had resectable biliary malignancy
* The patients who had hilar obstruction
* The patients who had duodenal obstruction
* The patients who had International Normalized Ratio (INR)>1.5
* The patients who did not give informed consent
* The patients who had technically difficult structure for Endoscopic retrograde cholangiopancreatography (ERCP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Re-intervention rate | 12 months
  Evaluation in both arms of the re-intervention rate considered as any procedure needed for a new drainage of the biliary tree, endoscopic or percutaneous, to replace a dysfunctional stent.

SECONDARY OUTCOMES:
Evaluation of patency, migration and adverse events rate | 12 months
  evaluation of patency, migration and adverse events rate for each arm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bowlus CL, Olson KA, Gershwin ME. Evaluation of indeterminate biliary strictures. Nat Rev Gastroenterol Hepatol. 2016 Jan;13(1):28-37. doi: 10.1038/nrgastro.2015.182. Epub 2015 Nov 3. PMID 26526122
- [Result] Reisman Y, Gips CH, Lavelle SM, Wilson JH. Clinical presentation of (subclinical) jaundice--the Euricterus project in The Netherlands. United Dutch Hospitals and Euricterus Project Management Group. Hepatogastroenterology. 1996 Sep-Oct;43(11):1190-5. PMID 8908550
- [Result] Zorron Pu L, de Moura EG, Bernardo WM, Baracat FI, Mendonca EQ, Kondo A, Luz GO, Furuya Junior CK, Artifon EL. Endoscopic stenting for inoperable malignant biliary obstruction: A systematic review and meta-analysis. World J Gastroenterol. 2015 Dec 21;21(47):13374-85. doi: 10.3748/wjg.v21.i47.13374. PMID 26715823
- [Result] Dumonceau JM, Tringali A, Papanikolaou IS, Blero D, Mangiavillano B, Schmidt A, Vanbiervliet G, Costamagna G, Deviere J, Garcia-Cano J, Gyokeres T, Hassan C, Prat F, Siersema PD, van Hooft JE. Endoscopic biliary stenting: indications, choice of stents, and results: European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline - Updated October 2017. Endoscopy. 2018 Sep;50(9):910-930. doi: 10.1055/a-0659-9864. Epub 2018 Aug 7. PMID 30086596
- [Result] Crippa S, Cirocchi R, Partelli S, Petrone MC, Muffatti F, Renzi C, Falconi M, Arcidiacono PG. Systematic review and meta-analysis of metal versus plastic stents for preoperative biliary drainage in resectable periampullary or pancreatic head tumors. Eur J Surg Oncol. 2016 Sep;42(9):1278-85. doi: 10.1016/j.ejso.2016.05.001. Epub 2016 May 24. PMID 27296728
- [Result] Mukai T, Yasuda I, Nakashima M, Doi S, Iwashita T, Iwata K, Kato T, Tomita E, Moriwaki H. Metallic stents are more efficacious than plastic stents in unresectable malignant hilar biliary strictures: a randomized controlled trial. J Hepatobiliary Pancreat Sci. 2013 Feb;20(2):214-22. doi: 10.1007/s00534-012-0508-8. PMID 22415652
- [Result] Tsuboi T, Sasaki T, Serikawa M, Ishii Y, Mouri T, Shimizu A, Kurihara K, Tatsukawa Y, Miyaki E, Kawamura R, Tsushima K, Murakami Y, Uemura K, Chayama K. Preoperative Biliary Drainage in Cases of Borderline Resectable Pancreatic Cancer Treated with Neoadjuvant Chemotherapy and Surgery. Gastroenterol Res Pract. 2016;2016:7968201. doi: 10.1155/2016/7968201. Epub 2016 Jan 6. PMID 26880897
- [Result] Yang MJ, Kim JH, Yoo BM, Hwang JC, Yoo JH, Lee KS, Kang JK, Kim SS, Lim SG, Shin SJ, Cheong JY, Lee KM, Lee KJ, Cho SW. Partially covered versus uncovered self-expandable nitinol stents with anti-migration properties for the palliation of malignant distal biliary obstruction: A randomized controlled trial. Scand J Gastroenterol. 2015;50(12):1490-9. doi: 10.3109/00365521.2015.1057219. Epub 2015 Jul 1. PMID 26133200
- [Result] Kitano M, Yamashita Y, Tanaka K, Konishi H, Yazumi S, Nakai Y, Nishiyama O, Uehara H, Mitoro A, Sanuki T, Takaoka M, Koshitani T, Arisaka Y, Shiba M, Hoki N, Sato H, Sasaki Y, Sato M, Hasegawa K, Kawabata H, Okabe Y, Mukai H. Covered self-expandable metal stents with an anti-migration system improve patency duration without increased complications compared with uncovered stents for distal biliary obstruction caused by pancreatic carcinoma: a randomized multicenter trial. Am J Gastroenterol. 2013 Nov;108(11):1713-22. doi: 10.1038/ajg.2013.305. Epub 2013 Sep 17. PMID 24042190
- [Result] Dumonceau JM, Kapral C, Aabakken L, Papanikolaou IS, Tringali A, Vanbiervliet G, Beyna T, Dinis-Ribeiro M, Hritz I, Mariani A, Paspatis G, Radaelli F, Lakhtakia S, Veitch AM, van Hooft JE. ERCP-related adverse events: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2020 Feb;52(2):127-149. doi: 10.1055/a-1075-4080. Epub 2019 Dec 20. PMID 31863440